CLINICAL TRIAL: NCT07245095
Title: Randomized Controlled Trial to Evaluate the Effect of Premedication With N-acetylcysteine and Simethicone on Mucosal Visibility During Elective Upper Gastrointestinal Endoscopy Using the TUGS Score
Brief Title: Premedication With N-acetylcysteine and Simethicone to Improve Mucosal Visualization in Elective Upper Endoscopy
Acronym: NACSIMET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital General de Mexicali (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: NACSIMET-ETDA-MEX2025
Record Dates: First submitted 2025-09-10; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Esophagogastroduodenoscopy; Simethicone; N-Acetylcysteine; Premedication; Visualization; Esophagogastroduodensocopy (EGD) Procedure; Placebo - Control; Gastritis Associated With Helicobacter Pylori; Tumor Gastric; Lesions in the Esophagus, Stomach, Duodenum or Rectum
Keywords: Esophagogastroduodenoscopy; Mucous Membrane; Premedication; Simethicone; Acetylcysteine; Gastrointestinal Tract
MeSH Terms: conditions — Stomach Neoplasms | interventions — Premedication; Acetylcysteine; Drinking Water; Simethicone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients receiving n-acetylcysteine/simethicone (Active Comparator)
  Interventions: Drug: Premedication with n-acetylcysteine; Drug: Premedication with simethicone
- Patients receiving placebo (Placebo Comparator)
  Interventions: Drug: Placebo (drinking water)

INTERVENTIONS:
Drug: Premedication with n-acetylcysteine — Once the sample size has been calculated, patients who meet the inclusion criteria will be recruited. who will be randomized using the "Randomized for Clinical Trial" program for assignment to treatment groups A and B. Group A will receive 600 mg of N-acetylcysteine and 100 mg of simethicone orally 20 to 60 minutes before the procedure, while the control group will receive an equivalent placebo infusion (composed of drinking water). Premedication and placebo will be labeled in containers as medication or placebo by external personnel not involved in the study, and the identification of each bag will be noted on a sheet and kept in an envelope that will be opened at the end of the study. Tolerance will be evaluated. If any adverse events are identified, the principal investigator will be notified for action regarding the management of the adverse event and its reporting.
  Arms: Patients receiving n-acetylcysteine/simethicone
Drug: Placebo (drinking water) — The control group will receive an equivalent placebo infusion (composed of drinking water)
  Arms: Patients receiving placebo
Drug: Premedication with simethicone — Once the sample size has been calculated, patients who meet the inclusion criteria will be recruited. who will be randomized using the "Randomized for Clinical Trial" program for assignment to treatment groups A and B. Group A will receive 600 mg of N-acetylcysteine and 100 mg of simethicone orally 20 to 60 minutes before the procedure, while the control group will receive an equivalent placebo infusion (composed of drinking water). Premedication and placebo will be labeled in containers as medication or placebo by external personnel not involved in the study, and the identification of each bag will be noted on a sheet and kept in an envelope that will be opened at the end of the study. Tolerance will be evaluated. If any adverse events are identified, the principal investigator will be notified for action regarding the management of the adverse event and its reporting
  Arms: Patients receiving n-acetylcysteine/simethicone

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled clinical trial is to assess whether the combination of N-acetylcysteine and simethicone improves mucosal visibility during upper gastrointestinal endoscopy in adults aged 18 to 99 years of both sexes, including both healthy individuals and those with non-bleeding gastrointestinal symptoms.

The main questions this study aims to answer are:

Does pre-endoscopy administration of N-acetylcysteine/simethicone improve mucosal visualization based on the Toronto Upper Gastrointestinal Cleanliness Score (TUGS)?

Is this combination safe and well tolerated in this patient population?

Researchers will compare patients receiving N-acetylcysteine (600 mg) and simethicone (100 mg) orally 20-60 minutes before the procedure with those receiving placebo (water) to determine if there is a significant improvement in TUGS scores.

Participants will:

Receive a single oral dose of either N-acetylcysteine/simethicone or placebo prior to endoscopy

Undergo a routine upper GI endoscopy

Have mucosal cleanliness evaluated using the TUGS scoring system

Be monitored for any adverse events or intolerance

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter clinical trial designed to evaluate the efficacy of N-acetylcysteine (NAC) combined with simethicone in improving mucosal visibility during upper gastrointestinal endoscopy (UGIE). The evaluation will be based on the Toronto Upper Gastrointestinal Cleanliness Score (TUGS), a validated tool to assess mucosal cleanliness.

Participants will include adult patients aged 18 to 99 years who are scheduled to undergo diagnostic UGIE for various indications and who do not present with active gastrointestinal bleeding. Eligible participants will be randomized to receive either a single dose of NAC (600 mg) plus simethicone (100 mg) or a placebo (water), administered orally 20 to 60 minutes prior to the procedure. The allocation will be blinded to both participants and endoscopists.

The main objective of the study is to determine whether this premedication protocol results in better mucosal visibility, as measured by the total TUGS score. Secondary objectives include documenting the presence of significant endoscopic findings and histopathological diagnoses, and evaluating the tolerability and safety profile of the premedication.

TUGS scores will be assigned by trained endoscopists blinded to the treatment allocation. Variables such as age, sex, BMI, duration of fasting, hospital site, and endoscope model will be recorded and controlled for in statistical analyses. The study will also assess any potential adverse events associated with the administration of NAC/simethicone.

This study is categorized as Phase 2 because it evaluates the preliminary efficacy and short-term safety of pre-procedural oral N-acetylcysteine (NAC) and simethicone to improve mucosal visibility during diagnostic upper gastrointestinal endoscopy, using the Toronto Upper Gastrointestinal Cleaning Score (TUGCS) as a validated surrogate endpoint. Both agents have established safety profiles for other indications, but their combined use for this indication is not an approved or established standard of care. The trial is randomized, double-blind, placebo-controlled with a moderate sample size designed to estimate effect size and variability rather than to deliver definitive, multi-center confirmatory evidence on hard clinical outcomes.

All procedures will adhere to ethical standards, and informed consent will be obtained from all participants. Data will be collected in a coded, anonymized format and analyzed using appropriate statistical methods, including ANCOVA and non-parametric tests where assumptions of normality are not met.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 70 years old.
* Patients who agree to participate in the clinical trial.
* Patients without active gastrointestinal bleeding.
* Signing of informed consent form.

Exclusion Criteria:

* Patients with a history of hypersensitivity to N-acetylcysteine
* Patients with a history of hypersensitivity to simethicone
* Patients with a previous endoscopic diagnosis
* Patients with a history of gastric or bariatric surgery
* Patients with a history of motor disorders (e.g., scleroderma, diabetic gastroparesis)
* Patients taking medications that delay gastric emptying (GLP-1 analogues)
* Pregnant or breastfeeding patients
* Patients who do not agree to participate in the clinical trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total score on the Toronto Upper Gastrointestinal Cleaning Score (TUGCS) | During the index upper endoscopy (Day 0), scored intra-procedure (≈20-60 minutes after premedication).
  The Toronto Upper Gastrointestinal Cleaning Score (TUGCS) is a validated scale that assesses mucosal cleanliness/visualization across four upper GI areas (fundus, body, antrum, and duodenum). Each area is scored from 0 to 3 (0 = poorest visualization; 3 = entire mucosa visible without suctioning/washing). The total score is the sum of all four areas (range 0-12). Higher scores indicate better mucosal cleanliness/visibility. Scoring is performed by blinded assessors during the procedure using standardized criteria.

SECONDARY OUTCOMES:
Detection of Mucosal Lesions | During endoscopy procedure
  Number of patients in whom mucosal lesions are detected during the procedure.
Complete Esophageal Visualization | During endoscopy.
  Binary assessment (Yes/No) of whether complete esophageal visualization was achieved.
Histological gastritis according to the Updated Sydney System (0-3 per item) and OLGA/OLGIM staging (0-IV) | Biopsies obtained during the index endoscopy (Day 0); histopathological report within 14 days
  Measurement tool: Updated Sydney System (sum of domains not mandatory).
  Sites and technique: 5 gastric biopsies according to the Sydney protocol (2 antrum, 2 body, 1 incisura angularis), fixed in formalin; H&E and Giemsa staining (or IHC if necessary for H. pylori).
  Domains and ranges (each 0-3):
  H. pylori density: 0 = absent, 1 = mild, 2 = moderate, 3 = marked.
  Chronic inflammation (mononuclear): 0-3.
  Activity (neutrophils): 0-3.
  Glandular atrophy: 0-3.
  Intestinal metaplasia: 0-3. Minimum-maximum range per domain: 0-3; higher scores = worse histological severity.
  Risk staging:
  OLGA (0-IV) for atrophy, OLGIM (0-IV) for intestinal metaplasia; higher stages = worse stage/higher risk.
  Reported measure: distribution of scores per domain (0-3) and proportion per OLGA/OLGIM stage (0-IV), comparing arms.
Presence and density of Helicobacter pylori by histology (Updated Sydney System 0-3) | Biopsies obtained during the index endoscopy (Day 0); report within 14 days
  Measurement tool: Updated Sydney System for H. pylori.
  Range and direction: 0-3 (0 = not detected; 1 = mild; 2 = moderate; 3 = marked). Higher scores = higher bacterial density.
  Technique: H&E + Giemsa staining (or IHC if indeterminate).
  Reported measure:
  Proportion of patients positive for H. pylori (≥1 on the scale), and
  Distribution of categories 0-3 per arm.
Number of histologically confirmed neoplasic lesions per patient | During the index endoscopy (Day 0) and histological confirmation up to 14 days
  Higher values reflect higher detection performance; this should be interpreted in conjunction with the detection rate (NDR)

CONTACTS AND LOCATIONS:
Locations (2):
- Mexico (2):
  - Hospital Almater, Mexicali, Estado de Baja California
  - Hospital General de Mexicali, Mexicali, Estado de Baja California

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data related to baseline demographics, Toronto Upper Gastrointestinal Cleaning Score (TUGS), endoscopic findings, and histopathological results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available beginning 6 months after publication of the main results and for up to 3 years thereafter.
Access Criteria: Researchers whose proposed use of the data has been approved by the study's principal investigator.

REFERENCES:
- [Background] Devereaux BM, Taylor ACF, Athan E, Wallis DJ, Brown RR, Greig SM, Bailey FK, Vickery K, Wardle E, Jones DM. Simethicone use during gastrointestinal endoscopy: Position statement of the Gastroenterological Society of Australia. J Gastroenterol Hepatol. 2019 Dec;34(12):2086-2089. doi: 10.1111/jgh.14757. Epub 2019 Jul 28. PMID 31242327
- [Background] Manfredi G, Berte R, Iiritano E, Alicante S, Londoni C, Brambilla G, Romeo S, Menozzi F, Griffanti P, Brandi G, Moreschi O, Pezzilli R, Zullo A, Buscarini E. Premedication with simethicone and N-acetylcysteine for improving mucosal visibility during upper gastrointestinal endoscopy in a Western population. Endosc Int Open. 2021 Feb;9(2):E190-E194. doi: 10.1055/a-1315-0114. Epub 2021 Jan 25. PMID 33532557
- [Background] Monrroy H, Vargas JI, Glasinovic E, Candia R, Azua E, Galvez C, Rojas C, Cabrera N, Vidaurre J, Alvarez N, Gonzalez J, Espino A, Gonzalez R, Parra-Blanco A. Use of N-acetylcysteine plus simethicone to improve mucosal visibility during upper GI endoscopy: a double-blind, randomized controlled trial. Gastrointest Endosc. 2018 Apr;87(4):986-993. doi: 10.1016/j.gie.2017.10.005. Epub 2017 Oct 14. PMID 29037773
- [Background] Beaufort IN, Verbeek RE, Bosman JH, Al-Toma A, Bogte A, Alvarez Herrero L, Weusten BLAM. Optimal timing of simethicone administration prior to upper endoscopy: A multicenter, single-blind, randomized controlled trial. Endosc Int Open. 2023 Oct 17;11(10):E992-E1000. doi: 10.1055/a-2157-5034. eCollection 2023 Oct. PMID 37854124
- [Result] Mahawongkajit P, Kanlerd A. A prospective randomized controlled trial comparing simethicone, N-acetylcysteine, sodium bicarbonate and peppermint for visualization in upper gastrointestinal endoscopy. Surg Endosc. 2021 Jan;35(1):303-308. doi: 10.1007/s00464-020-07397-8. Epub 2020 Feb 3. PMID 32016519
- [Result] Chang WK, Yeh MK, Hsu HC, Chen HW, Hu MK. Efficacy of simethicone and N-acetylcysteine as premedication in improving visibility during upper endoscopy. J Gastroenterol Hepatol. 2014 Apr;29(4):769-74. doi: 10.1111/jgh.12487. PMID 24325147
- [Result] Sajid MS, Rehman S, Chedgy F, Singh KK. Improving the mucosal visualization at gastroscopy: a systematic review and meta-analysis of randomized, controlled trials reporting the role of Simethicone +/- N-acetylcysteine. Transl Gastroenterol Hepatol. 2018 May 19;3:29. doi: 10.21037/tgh.2018.05.02. eCollection 2018. PMID 29971260
- [Result] Li Y, Du F, Fu D. The effect of using simethicone with or without N-acetylcysteine before gastroscopy: A meta-analysis and systemic review. Saudi J Gastroenterol. 2019 Jul-Aug;25(4):218-228. doi: 10.4103/sjg.SJG_538_18. PMID 31044749